CLINICAL TRIAL: NCT05754216
Title: Intraoperative Identification and Stimulation of the Glossopharyngeal Nerve
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants have been enrolled to date.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Kent, Associate Professor, Department of Otolaryngology-Head and Neck Surgery, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 230171
Record Dates: First submitted 2023-02-13; First posted 2023-03-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Obstructive Sleep Apnea
MeSH Terms: conditions — Head and Neck Neoplasms; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All patients who meet eligibility will undergo a planned resection of parapharyngeal space (PPS) mass for management of head and neck cancer and will have measurements and photos/videos of the common trunks taken. Fine-wire electrodes will be placed on these nerve branches. For each patient, if the target nerve branches can be identified and electrodes successfully placed, they will additionally undergo drug-induced sleep endoscopy (DISE) immediately following PPS surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surgical Procedure (Other): Consented patients who meet eligibility will have a surgical procedure for management of head and neck cancer, with dissection and exposure of the relevant anatomic structures as part of regular clinical care.
  Interventions: Device: Nerve stimulation using nerve stimulation device and sterile wire electrode.

INTERVENTIONS:
Device: Nerve stimulation using nerve stimulation device and sterile wire electrode. — A nerve stimulator device will be used in this study as a research tool to investigate whether a future (currently nonexistent) medical device might be able to stimulate desired pharyngeal musculature in a therapeutic manner.

SUMMARY:
Published data suggest that the glossopharyngeal nerve innervates pharyngeal musculature important for maintenance of upper airway patency. The investigators propose a study examining the anatomic variation of the glossopharyngeal nerve and the effect of electrical stimulation on muscle recruitment and upper airway patency.

DETAILED DESCRIPTION:
This is a single-arm physiology study. Consenting patients undergoing parapharyngeal space (PPS) surgery for tumor extirpation will undergo dissection of the glossopharyngeal nerve branches to the stylopharyngeus and pharyngeal constrictor muscles. Fine-wire electrodes will be placed on these nerve branches. For each patient, if the target nerve branches can be identified and electrodes successfully placed, they will additionally undergo drug-induced sleep endoscopy (DISE) immediately following PPS surgery.

Per routine care, an incision is made across the neck to provide surgeons access to parapharyngeal space for tumor extirpation. During this dissection, the branch(es) of the glossopharyngeal nerve innervating the stylopharyngeus (SP) and pharyngeal constrictor (PC) muscles are exposed. For this study, measurements and photos/videos of the nerve will be taken. A fine-wire electrode will be placed on either or both successfully identified nerves and stimulated to assess muscle activation and changes in upper airway patency.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults with BMI ≥ 25 and ≤ 40 kg/m2
* Planned resection of parapharyngeal space (PPS) mass without clinical evidence of cranial nerve function deficits based on physical examination
* History of moderate-to-severe Obstructive Sleep Apnea (OSA) as confirmed by previous polysomnogram OR high risk for OSA based on STOP-BANG criteria (STOP-BANG score ≥ 3)

Exclusion Criteria:

* Unable to consent for research due to a pre-existing neurologic condition or language barriers as determined by PI
* History of other primary sleep-related breathing disorder (e.g., central, or complex sleep apnea).
* Previous pharyngeal surgery excluding tonsillectomy (e.g. cleft palate repair, uvulopalatopharyngoplasty)
* Prior history of head and/or neck chemoradiation therapy
* Existing indwelling neurostimulation device (e.g. pacemaker; spinal, vagal, or hypoglossal nerve stimulator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in variation in the conformation of the glossopharyngeal nerve | Collected during a single operative procedure, taking about 15 minutes.
  The natural variation in the conformation of the glossopharyngeal nerve will be measured by length, diameter, and conformation of the common trunk and its dependent branches to the Stylopharyngeus Muscle (SP) and Pharyngeal Constrictor Muscles (PC), measured in mm with a flexible ruler.

SECONDARY OUTCOMES:
Change in Airway cross-sectional diameter | Collected during a single DISE procedure, taking about 15 minutes.
  Change in airway cross-sectional diameter will be measured throughout the operative procedure via flexible fiberoptic nasopharyngoscopy.
Change in airflow | Collected during a single DISE procedure, taking about 15 minutes.
  Airflow (L/min) will be measured throughout the operative procedure via a pneumotachometer applied to the nose.
Change in upper airway pressure | Collected during a single DISE procedure, taking about 15 minutes.
  Upper airway pressure changes (cmH20) will be measured throughout the operative procedure via a pneumotachometer applied to the nose.
Change in respiratory effort | Collected during a single DISE procedure, taking about 15 minutes.
  Respiratory effort data (mV) will be measured throughout the operative procedure via two respiratory inductance plethysmography belts.

CONTACTS AND LOCATIONS:
Overall Officials: David T. Kent, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No